CLINICAL TRIAL: NCT05336162
Title: Retention Rate and Caries Preventive Effect of Self Etch Giomer Based Fissure Sealant Versus Total Etch Resin Based Fissure Sealant in Patients With Non- Cavitated Pits and Fissures in Permanent Molars Over One Year.
Brief Title: Retention Rate and Caries Preventive Effect of Self Etch Giomer Based Fissure Sealant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Radwa Wael Maher, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: giomer based fissure sealant
Record Dates: First submitted 2022-04-08; First posted 2022-04-20 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Fissure Sealant

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with non-cavitated pits and fissures in permanent molars will be treated with BeautiSealant (Experimental): Young adults (16-22 y) who have existing pits and fissures that are anatomically deep and caries susceptible or with Stained pits and fissures with minimum decalcification of opacification and no softness at the base of the fissure (ICDAS 1 and 2).
  Interventions: Other: Self etch giomer based fissure sealant (BeautiSealant, Shoufu, USA)
- Patients with non-cavitated pits and fissures in permanent molars will be treated with UltraSeal XT (Active Comparator): Young adults (16-22 y) who have existing pits and fissures that are anatomically deep and caries susceptible or with Stained pits and fissures with minimum decalcification of opacification and no softness at the base of the fissure (ICDAS 1 and 2).
  Interventions: Other: Self etch giomer based fissure sealant (BeautiSealant, Shoufu, USA)

INTERVENTIONS:
Other: Self etch giomer based fissure sealant (BeautiSealant, Shoufu, USA) — A fissure sealant providing a physical barrier that inhibits microorganisms and food particles accumulation, preventing caries initiation, and arresting caries progression

SUMMARY:
With limited evidence-based information in literature about using giomer based pit and fissure sealant(BeautiSealant) in non-cavitated pits and fissures in permanent molars, it is beneficial to evaluate the newly introduced material using a randomized controlled clinical trial to test the null hypothesis that this new pit and fissure sealant (BeautiSealant, Shoufu, USA). will have the same effect as resin based pit and fissure sealant (UltraSeal XT™ plus, Ultradent, USA) regarding retention rate and caries preventive effect.

DETAILED DESCRIPTION:
Giomer is an adhesive material in dentistry made from resin that contains a Pre-Reacted Glass- ionomer (PRG) filler. The advantages of Giomer include the release and recharge of fluoride, resistance to acid, anti-plaque effect, remineralization of dentin, and acid buffering capacity. The surface pre-reacted glass-ionomer filler containing sealant (BeautiSealant) demonstrated superior fluoride recharging properties. BeautiSealant is filled with Shofu's proprietary S-PRG (Surface Pre-Reacted Glass) with cariostatic properties, acid neutralization, and plaque inhibition decreasing the risk for secondary caries. Beautisealant unlike traditional sealants which require phosphoric acid etching, demineralizing and dehydrating healthy teeth, shoufu's self etching primer is significantly less acidic helping to preserve healthy tooth structure and still maintaining equal or better shear bond strength. The clinical use of self-etching agents could be recommended before pit and fissure sealants application in new dental protocols. No clinical trials have been published uptill now evaluating caries incidence around giomer based fissure sealant by VistaCam iX proof. The aim of this study is to Evaluate the retention rate of self etch giomer based fissure sealant and also caries incidence using VistaCamiX.

ELIGIBILITY:
Inclusion Criteria:

* Young adults (16-22 y).
* Patients who have existing pits and fissures that are anatomically deep and caries susceptible.
* Permanent molars teeth without any caries and cavitation.
* Permanent molar teeth that have deep pit and fissure morphology, with "sticky" fissures. •Permanent molar teeth with stained grooves.
* Stained pits and fissures with minimum decalcification of opacification and no softness at the base of the fissure (ICDAS 1 and 2).

Exclusion Criteria:

* Uncooperative behavior, limits the use of sealants due to hampering of adequate field or isolation techniques throughout the procedure.
* Patients allergic to sealant material.
* Patient with history of medical disease, drug therapies or any other serious relevant problem.
* An individual with no previous caries experience and well coalesced pits and fissures
* Partially erupted teeth.
* Teeth with cavitation or caries of the dentin.
* A large restoration is present on occlusal Surface.
* If pits and fissures are self-cleansable.
* Teeth with dental fluorosis, hypocalcification or hyper calcification.

Ages: 16 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2024-01-25 (Estimated); Study Completion 2024-06-25 (Estimated)

PRIMARY OUTCOMES:
Retention Rate of sealant | 12 months
  1-Full retention: the materials were fully present on the occlusal surfaces. 2- Partially lost: the materials were present, but as a result of either wear or loss of the material, part of a previously sealed pit or fissure, or both, was exposed. 3-Totally lost: no trace of materials was detected on the surface.

SECONDARY OUTCOMES:
Caries Incidence | T0=Baseline immediate postoperative. T1= 3 months follow up. T2= 6 months follow up. T3=12 months follow
  Intra-oral fluorescence camera VistaCamiX proof camera using (Software Program)

CONTACTS AND LOCATIONS:
Locations (1):
- Radwa Wael, Cairo, Egypt